CLINICAL TRIAL: NCT07334977
Title: Synergistic Potential of Non-invasive Brain and Spinal Cord Stimulation for Improving Sensorimotor and Cognitive Functions After Neurological Injury
Brief Title: Synergistic Effect of Non-invasive Brain and Spinal Cord Stimulation
Acronym: BrainSpineStim
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre National de la Recherche Scientifique, France (Other)
Collaborators: University Hospital, Bordeaux (Other); Centre de la Tour de Gassies (Unknown); Institute of Neurodegenerative Diseases, CNRS UMR 5293 (Unknown)
Responsible Party: Principal Investigator, Fabien Wagner, Principal investigator, Centre National de la Recherche Scientifique, France
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-A00724-43; ARF202309017508 (Other Grant/Funding Number: Fondation pour la Recherche Médicale)
Record Dates: First submitted 2025-08-28; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Spinal Cord Injury; Able Bodied
Keywords: Neuromodulation; Neuroplasticity; transcutaneous Spinal Cord Stimulation; transcranial Direct Current Stimulation; Neuroimaging
MeSH Terms: conditions — Stroke; Spinal Cord Injuries | interventions — Transcranial Direct Current Stimulation; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- tDCS+CMT (Experimental): tDCS administered during the performance of cognitive and motor task for 20 min
  Interventions: Procedure: tDCS; Behavioral: Cognitive-Motor Task
- tSCS+CMT (Experimental): 20-min tSCS administered during the performance of cognitive and motor task for 20 min
  Interventions: Procedure: tSCS; Procedure: Sham
- tDCS-tSCS+CMT (Active Comparator): tDCS associated with tSCS administered during the performance of cognitive and motor task for 20 min
  Interventions: Procedure: tDCS; Procedure: tSCS; Behavioral: Cognitive-Motor Task
- Sham-tDCS-tSCS+CMT (Sham Comparator): Sham tDCS associated with Sham tSCS administered during the performance of cognitive and motor task for 20 min
  Interventions: Procedure: tDCS; Procedure: tSCS; Procedure: Sham; Behavioral: Cognitive-Motor Task

INTERVENTIONS:
Procedure: tDCS — tDCS will be delivered using an electrical stimulation device d (1X1 tES, Soterix Medical Inc., USA, CE marked) delivering a direct current at 2 mA for a period of 20 minutes. Silicone electrodes are placed in sponges soaked in physiological saline (5 cm × 7 cm) (EASYpadTM, Soterix Medical Inc.), with the anode and cathode centered on the optimal cortical areas determined during testing visits.
  Other Names: transcranial Direct Current Stimulation
  Arms: Sham-tDCS-tSCS+CMT; tDCS+CMT; tDCS-tSCS+CMT
Procedure: tSCS — tSCS will be applied for 20 minutes using a constant current electrical stimulator (DS5 or DS7A, Digitimer Ltd, CE marked) delivering monophasic pulses at 30 Hz at stimulation sites and intensities specific to each participant and defined in advance during testing visits.
  Other Names: transcutaneous Spinal Cord Stimulation
  Arms: Sham-tDCS-tSCS+CMT; tDCS-tSCS+CMT; tSCS+CMT
Procedure: Sham — For the sham stimulation interventions, the current slowly increases to the intensity used during the active interventions for 30 seconds, then slowly decreases over the next 30 seconds, at the beginning and end of the stimulation. The sham interventions use the same electrode placements as during the active ones for a total duration of 20 min.
  Arms: Sham-tDCS-tSCS+CMT; tSCS+CMT
Behavioral: Cognitive-Motor Task — The cognitive-motor task will be administered using the ArmeoControl software supplied with the ArmeoSping® or ArmeoPower® upper limb rehabilitation exoskeleton. Participants will be seated in a chair or their wheelchair and fitted into the exoskeleton.The exoskeleton is linked to a series of exercises performed on a computer via a virtual reality interface (ArmeoControl), which allows simultaneous training of the arms and hands in a large workspace. Two vertical and horizontal "visually guided reaching" tasks will be offered, each lasting 10 minutes. These tasks are chosen to provide training in cognitive-motor functions (grabbing a target moving in a virtual workspace) and sensorimotor functions (interacting with the exoskeleton to move the target).
  Arms: Sham-tDCS-tSCS+CMT; tDCS+CMT; tDCS-tSCS+CMT

SUMMARY:
The goal of this clinical study is to investigate the potential synergy between non-invasive brain and spinal cord stimulation administered during a cognitive-motor task, in terms of their immediate effects on sensorimotor and cognitive functions after neurological injuries affecting the upper limb (cervical spinal cord injury and stroke). Secondary objectives are to evaluate the relevance of anatomical MRI, functional MRI, and neurophysiological measurements for optimizing and predicting the effects of these different interventions.

DETAILED DESCRIPTION:
Over the past decade, innovative electrical stimulation strategies have emerged to improve the effectiveness of conventional rehabilitation approaches following spinal cord injury or stroke. Transcranial direct current stimulation (tDCS) and transcutaneous spinal cord stimulation (tSCS) are two non-invasive stimulation techniques targeting respectively the brain and spinal cord. These techniques have demonstrated immediate and lasting positive effects on the recovery of lost neurological functions following damage to the brain (in the case of stroke) or the spinal cord (in the case of spinal cord injury). Functional improvements leading to a better quality of life have been demonstrated in response to tSCS or tDCS sessions combined with motor training. Recent studies suggest a potential synergistic effect of these two types of intervention, which we propose to characterize in control participants, participants with cervical spinal cord injury, and post-stroke participants.

OBJECTIVES: In this project, we seek to study the potential synergistic effects of an intervention combining non-invasive stimulation of the brain and spinal cord, administered during the performance of a cognitive-motor task, compared to a control intervention and each intervention administered separately, on the recovery of motor and cognitive-motor functions after neurological injury. Secondary objectives are to evaluate the relevance of anatomical MRI data and neurophysiological measurements for optimizing and predicting the effects of these different interventions.

METHODOLOGY/RESEARCH DESIGN: Single-center, prospective, comparative, randomized, crossover, and single-blind clinical study comparing four neuromodulation interventions: S1: tDCS, S2: tSCS, S3: tDCS-tSCS, S4: sham, administered during a cognitive-motor training task of the affected upper limb using the Armeo technology. Three groups of participants will be included: one control group, one group with cervical spinal cord injury, and one post-stroke group. The two groups with either spinal cord injury or stroke will participate in a total of nine visits: the inclusion visit, four testing visits, and four intervention visits. The control group will participate only in the inclusion and testing visits. Outcome measures will include neurophysiological and clinical performance measures.

ELIGIBILITY:
Inclusion Criteria:

CONTROL GROUP:

* Over 18 years of age
* Participant who has signed an informed consent form
* Participant who is affiliated with and covered by the social security system

POST-STROKE GROUP:

* Over 18 years of age
* Who sustained a stroke more than 3 weeks ago
* Considered medically stable by the medical investigator
* Who has signed an informed consent form
* Affiliated with and covered by the social security system

SCI GROUP:

* Over 18 years of age
* Considered to have a complete or incomplete spinal cord injury (i.e., with a score on the Spinal Injury Association (ASIA) Impairment Scale (AIS) score from A to D)
* Considered medically stable by the investigating physician
* Presenting with quadriplegia due to cervical injury
* Who has signed an informed consent form
* Affiliated with and covered by the social security system.

Exclusion Criteria:

* Suffering from a chronic condition
* Skin problems or open wounds
* History of epilepsy or seizures
* Presence of a contraindication to the use of magnetic/electrical stimulation or MRI, including: cardiac pacemaker; implanted hearing aid; intraocular foreign body, shrapnel, or bullets; metal worker; pacemaker or neurostimulator; claustrophobia
* Presence of implanted medical devices (cardiac valve, endovascular devices, ventricular shunt valve, surgical clips, metallic sutures, staples, stent, osteosynthesis or arthrodesis hardware) not classified as "MR Conditional" according to ASTM F2503.
* Individuals who are legally incompetent, under judicial protection, guardianship, or trusteeship
* Pregnant and/or breastfeeding women
* Individuals who refuse to be informed of any abnormalities that may be detected by MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Sensory Performance | Immediately post-intervention at interventional visits 1, 2, 3, and 4 (days 14, 18, 21, 25)
  GRASSP subscores: Hand dorsal and palmar sensory function
Quantitative Prehension Performance | Immediately post-intervention at interventional visits 1, 2, 3, and 4 (days 14, 18, 21, 25)
  GRASSP Quantitative Prehension Subscore: Hand prehension motor performance

SECONDARY OUTCOMES:
Cognitive performance | Immediately post-intervention at interventional visits 1, 2, 3, and 4 (days 14, 18, 21, 25)
  Total score on the ECAS multi-domain assessment
Safety of the intervention | Immediately post-intervention at interventional visits 1, 2, 3, and 4 (days 14, 18, 21, 25)
  Safety questionnaire describing side effect appearance and their relative severity. The frequency of a specific side effect will be computed and the severity score (1 to 4) will be averaged across participant
Feasibility of the intervention | Immediately post-intervention at interventional visits 1, 2, 3, and 4 (days 14, 18, 21, 25)
  4-item instrument measuring the feasibility of an intervention. The total score is calculated by summing the four items, yielding a range from 4 to 20, with higher scores indicating greater perceived feasibility of the intervention.
Neurophysiological assessment of posterior root-muscle reflexes | Immediately post-intervention at testing visit #2 (day 4)
  Upper-limb electromyographic (EMG) responses during paired-pulse tSCS

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Wagner, PhD, Principal Investigator — Institute of Neurodegenerative Diseases, CNRS UMR 5293; Nabila Brihmat, PhD, Principal Investigator — Institute of Neurodegenerative Diseases, CNRS UMR 5293; Hélène Cassoudesalle, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - Service de Médecine Physique & Réadaptation - CHU Bordeaux, Bordeaux
  - Centre de la Tour de Gassies, Bruges

IPD SHARING:
Plan to Share IPD: Undecided
Based on request and on the data type requested and ethically approved (only non-personally Identifiable Information).